CLINICAL TRIAL: NCT04873115
Title: Double-blind, Placebo-controlled, Randomized Clinical Trial Comparing the Efficacy and Safety of Sialanar Plus orAl rehabiLitation Against Placebo Plus Oral Rehabilitation for chIldren and Adolescents With seVere Sialorrhoea and Neurodisabilties,
Acronym: SALIVA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Proveca Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO-GLY-002 / E2013
Record Dates: First submitted 2021-04-27; First posted 2021-05-05 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Sialorrhea; Neurodevelopmental Disorders
Keywords: Pediatric; sialorrhea; neurodisability
MeSH Terms: conditions — Sialorrhea; Neurodevelopmental Disorders | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Double-blinded randomised phase followed by open label treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sialanar (Active Comparator): Sialanar administered as per the SmPC - titration over 4 weeks to reach a dose balancing efficacy with tolerability.
  Interventions: Drug: Sialanar; Other: Oral Rehabilitation
- Placebo (Placebo Comparator): Placebo administered as per the Sialanar SmPC - titration over 4 weeks to reach a dose balancing efficacy with tolerability.
  Interventions: Other: Placebo; Other: Oral Rehabilitation

INTERVENTIONS:
Other: Placebo — Sialanar placebo
  Arms: Placebo
Drug: Sialanar — Sialanar - a licensed glycopyrronium bromide product
  Arms: Sialanar
Other: Oral Rehabilitation — Standard oral rehabilitation for provided drooling

SUMMARY:
Double blind, placebo-controlled, randomised trial, multicentre in France with open-label tolerability phase.

The double-blind placebo-controlled study duration will be scheduled for 3 months with the final visit of the double-blind period at D84. After the D84 assessment, patients will be invited to continue into a 6-month openlabel study extension (OLSE) with ex-Sialanar® patients continuing the treatment and ex-placebo patients starting Sialanar®

DETAILED DESCRIPTION:
This is a phase 4, double-blind, placebo-controlled, randomised trial, multicentre study conducted in France to evaluate the efficacy and safety of glycopyrronium bromide (Sialanar®) versus placebo in addition to Standard of Care (SOC) management (rehabilitation) in children with severe sialorrhea related to chronic neurodisabilities, i.e cerebral palsy, Angelman syndrome, Rett's syndrome, epilepsy, amyotrophic lateral sclerosis and mental retardation. The patient population will be children aged from 3 to 17-year-old with severe sialorrhea due to chronic neurological disorders, defined as a score of at least 6 on the modified Teachers Drooling Scale (mTDS), after at least 3 months of non pharmalogical rehabilitation. A total of 80 patients who meet the eligibility criteria (see section 6.3) will be enrolled in the study. General eligibility criteria will be assessed and the DIS scale (French validated version) performed at the enrolment visit. Patients, enrolled in the study, will be randomized to receive the study drug in a doubleblind fashion, either Sialanar® of placebo. Eligible patients will be randomized in a 1:1 ratio into the 2- treatment arms with no additional stratification. Patients will receive the study drug, an oral solution, 3 times daily during the 3-month blind period. The titration will be performed during the first 5 weeks as detailed in section 7.1.3 Outpatient visits will occur at D28 and D84. Telephone interviews will occur every week during the titration period and at D56.

The double-blind placebo-controlled study duration will be scheduled for 3 months with the final visit of the double-blind period at D84. After the D84 assessment, patients will be invited to continue into a 6-month open-label study extension (OLSE) with ex-Sialanar® patients continuing the treatment and ex-placebo patients starting Sialanar®. An period of titration will be performed for patients starting Sialanar®, monitored by weekly telephone interviews. Telephone interviews will also be scheduled at D140. Clinic visit will be scheduled at D168 for all patients. Final OLSE visit will occur at D252. Patients will be assessed for disease response with the Drooling Impact Scale (DIS) including 10 items rated on a scale from 1 to 10 at D0 and during follow-up visits at D28, D84 and D252. Quality of Life will be evaluated through the DISABKIDS self-reported instrument completed by parents/ caregivers as well as children, when possible. Adverse events will be collected at every visit from parent or carer and participant where possible. All adverse events will be recorded at every scheduled visit plus outside of visits as required. All SAEs and SUSARs will be recorded and reported as per standard EMA guidelines (cf. Section 9.2).

The duration of the study will approximately be 15 months including 6 months of enrolment and 9 months of follow up from the last patient enrolled (3 months for the blind period and 6 months for the OLSE). The end of the blind period will correspond to the last patient completed D84 visit. The end of the OLSE will correspond to the last patient completed D252 visit. After all patients complete the blind period, the final analysis of the primary outcome (change in DIS at D84) will be performed. The follow up analysis of the OLSE period will be carried after all patients ended the study. All safety data will be analysed regardless of the outcome of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged ≥ 3 years old and < 18 years old.
2. Children with weight ≥ 13 kg
3. Children with chronic neurological disorders (such as polyhandicap, cerebral palsy, Angelman syndrome, Rett's syndrome, epilepsy, amyotrophic lateral sclerosis and mental retardation)
4. Diagnosis of severe sialorrhoea due to a chronic neurological disorder as assessed by a modified Teachers Drooling Scale (mTDS) ≥ 6.
5. DIS Scale ≥ 50. Impact of drooling as assessed by drooling impact scale.
6. Children who have completed at least 3 months of non-pharmacological standard of care treatment (i.e. rehabilitation e.g. intraoral stimulation and oral facial exercise).
7. Children with stable drooling for the past 4 weeks.
8. Written consent form signed by parents (or, when applicable, the subject's legally acceptable representative).
9. Affiliated or beneficiary of a social security scheme.
10. A nominated parent or carer who can commit to complete parent / carer questionnaires, with good ability to understand and speak French.
11. Children testing negative for COVID-19 at start of the trial. (Asymptomatic children with a positive test have the opportunity to have a re-test at least 2 weeks following the initial test and must be negative on the re-test for inclusion).

Exclusion Criteria:

1. Children unwilling to provide assent to participate in the study. (children who are unable to provide assent should be considered eligible).
2. Botulinum injection for sialorrhoea given within 6 months of enrolment.
3. Any anticholinergic therapy used in the previous 4 weeks.
4. Scopoderm patch used in the previous 4 weeks.
5. History of surgery for drooling in the previous 12 months.
6. Children prescribed non-permitted concomitant medication as defined in section 7.2.2
7. Children in whom anticholinergics are contraindicated such as those with glaucoma, myasthenia gravis, urinary retention, severe renal impairment, history of intestinal obstruction, ulcerative colitis, paralytic ileus, pyloric stenosis or hypersensitivity to the active substance or the excipient.
8. On-going or programmed orthodontic treatment over the study period.
9. Untreated oro-mandibular dystonia (isolated lingual dystonia accepted), clinical gastro oesophageal reflux, dental inflammatory condition (dental caries, gingivitis…).
10. Family and carers unable to commit to the schedule of the study protocol.
11. Female patients who are lacting or pregnant
12. Female patients who are planning a pregnancy within the study period
13. Patients having participated in another clinical study within at least 30 days or within 5 half-lives of last dose of IMP (whichever is longer).
14. Patients receiving systemic immunosuppressive treatment including cyclosporin, methotrexate, azathioprine cyclophosphamide, mycophenolic acid, anti TNFα, monoclonal antibodies or with congenital immunodeficiency

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
The Change in Drooling Impact Scale (DIS) between baseline and D84. | 84 days
  DIS possible range is 10-100. Lower score indicates a better outcome.

SECONDARY OUTCOMES:
Change in Drooling Impact Scale (DIS) between baseline and D28. | 28 days
  DIS possible range is 10-100. Lower score indicates a better outcome.
Proportion of responders at D84 (a response is defined as a DIS improvement ≥ 13.6 points). | 84 days
  DIS possible range is 10-100. Lower score indicates a better outcome.
Proportion of responders at D28 (a response is defined as a DIS improvement ≥ 13.6 points). | 28 days
  DIS possible range is 10-100. Lower score indicates a better outcome.
Proportion of good responders at D84 (a good response is defined as a DIS improvement ≥ 28 points). | 84 days
  DIS possible range is 10-100. Lower score indicates a better outcome.
Changes in the number of used bibs or clothing over 7 days (Item 3 of the DIS) at D84 | 84 days
Changes in the number of used bibs or clothing over 7 days (Item 3 of the DIS) at D28 | 28 days

OTHER OUTCOMES:
Change in the DIS 10-point item 9 from baseline. "To what extent did your child's drooling affect his or her life?" to D28 and D84. | 28 and 84 days
  DIS possible range is 10-100. Lower score indicates a better outcome.
Change in in the DIS 10-point item 10 from baseline. "To what extent did your child's dribbling affect you and your family's life?" to D28 and D84. | 28 and 84 days
  DIS possible range is 10-100. Lower score indicates a better outcome.
The change in DISABKIDS instrument from baseline to D84. | 84 days
Adverse events recorded from baseline to day 84, including all AEs and SAE. | 84 days
Changes in DIS Scale between baseline and D252 and between D84 and D252 in the previous 'Sialanar®-arm' patients. | up to 252 days
  DIS possible range is 10-100. Lower score indicates a better outcome.
Change in DIS Scale between D84 and D252 for patients previously taking placebo | 168 days
  DIS possible range is 10-100. Lower score indicates a better outcome.
Change in the DIS 10-point item 9. "To what extent did your child's drooling affect his or her life?" between baseline and D252. | 252 days
  DIS question 9 possible range is 1-10. Lower score indicates a better outcome.
Change in the DIS 10-point item 10. "To what extent did your child's dribbling affect you and your family's life?" between baseline and D252. | 252 days
  DIS question 10 possible range is 1-10. Lower score indicates a better outcome.
Change in DISABKIDS instrument score between baseline and D252. | 252 days
Adverse events recorded from D84 to D252 | 168 days

CONTACTS AND LOCATIONS:
Overall Officials: Nick Probert, Study Director — Proveca Pharma Limited; Pierre Fayoux, Principal Investigator — CHU Lille
Locations (1):
- CHU Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No